CLINICAL TRIAL: NCT06904534
Title: Comparison of Fetal Cardiac Functions in Pregnant Women Using Nifedipine and Magnesium Sulfate for Tocolysis
Brief Title: Fetal Cardiac Effects of Tocolytic Nifedipine and Magnesium Sulfate
Status: Active, not recruiting | Type: Observational
Sponsor: Sanliurfa Education and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: SEAH-CARD
Record Dates: First submitted 2025-03-23; First posted 2025-04-01 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Unexpected Fetal Cardiac Effects of Nifedipine and MgSO4
Keywords: Nifedipine; MgSO4; Fetal echocardiography.

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pregnancies using nifedipine and MgSO4 for tocolytic purposes

SUMMARY:
The potential unexpected effects of nifedipine and MgSO4, the tocolytic agents used for the indication of preterm labor, on fetal heart will be determined. In this study, the fetal echocardiographic findings of nifedipine and MgSO4 will be compared.

DETAILED DESCRIPTION:
This study will include pregnancies at 24-34 weeks of gestation that are using nifedipine and MgSO4 for tocolysis. Fetal echocardiographic findings of these pregnancies will be recorded

ELIGIBILITY:
Inclusion Criteria:-Patients with preterm labor indication at 24-34 weeks of gestation

-Treated with nifedipine or MgSO4 for tocolysis

Exclusion Criteria:

* Multiple pregnancy
* premature rupture of membranes
* Chorioamnionitis
* Placental abruption
* Severe fetal growth restriction
* Congenital anomalies of the fetus
* Preeclampsia
* Oligohydramnios
* Maternal diabetes
* Contraindications for the use of nifedipine and/or MgSO4 in the mother

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Patients with preterm labor indication at 24-34 weeks of gestation who are treated with nifedipine or MgSO4 for tocolysis
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Use of nifedipine or MgSO4 as tocolytic agents | Fetal echocardiographic findings after 48 hours the use of nifedipine or MgSO4
  Pregnancies between 24-34 weeks of gestation using nifedipine and MgSO4 for tocolysis will be evaluated. Preterm labor is defined as persistent uterine contractions (at least two contractions every 10 minutes or four contractions in 1 hour) resulting in cervical changes (at least 80% effacement and 2 cm cervical dilation). Nifedipine will be administered as an initial 10 mg oral loading dose every 20 minutes for one hour, followed by 10 mg oral maintenance doses every 6 hours for 48 hours. The MgSO4 treatment protocol involves a 100 mL infusion of 5% dextrose containing 4-6 grams of MgSO4 (MgSO4 15% amp.) as an intravenous (IV) loading dose over 20 minutes, followed by a maintenance dose of 2 grams per hour IV. During treatment, patients will be monitored hourly for urination patterns, deep tendon reflexes, and respiratory rate. Treatment will be stopped 6 hours after the cessation of contractions. Doppler measurements will be taken before the first treatment dose and 48 hours after.

CONTACTS AND LOCATIONS:
Locations (1):
- Şanlıurfa Training and Research Hospital, Sanliurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No